CLINICAL TRIAL: NCT00729170
Title: Impact of Milk Supplementation on Body Composition, Bone Density and Satiety in Women Following a Weight Loss Program.
Brief Title: Milk Supplementation and Energy Balance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Dairy Farmers of Canada (Other); National Dairy Council (Other)
Responsible Party: Principal Investigator, Angelo Tremblay, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1_Tremblay
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Osteoporosis
Keywords: Milk; Calcium; Weight loss; Bone density; Appetite
MeSH Terms: conditions — Obesity; Osteoporosis; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Supplementation of milk (35% more calcium) — The supplement provides 1000 mg of calcium and 250 kcal daily.

SUMMARY:
The aim of the project is to determine if milk supplementation during a caloric restriction program facilitates the lost of weight, improves the appetite control and attenuates the decrease of bone mineral content in low-calcium consumer women.

DETAILED DESCRIPTION:
Calcium deficiency is related to a higher risk of obesity. Some studies showed a lost of weight by elevating the calcium consumption to reach the recommended level. Milk supplementation could be a good alternative to reach this objective, but its impact on weight loss and on appetite sensations has not been verified. Furthermore, losing weight leads to some negative consequences like a decrease of bone mineral content. Considering the benefits of milk on bone health, a higher intake of this food product during weight loss could represent a healthy strategy.

ELIGIBILITY:
Inclusion Criteria:

* Low-calcium consumer (less than 800 mg daily)
* BMI between 27 to 42 kg/m2
* Sedentary
* Healthy

Exclusion Criteria:

* In menopause
* Medications that alter the project's objectives
* Smoker
* Dietary supplement consumer
* High alcohol or caffeine consumer

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Body composition (body weight, fat mass, anthropometric measurements) | Baseline, month 1, and month 6

SECONDARY OUTCOMES:
Bone density (DXA) | Baseline and month 6
Appetite sensations | Baseline, month 1, and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Tremblay, Ph.D., Principal Investigator — Laval University; Denis R Joanisse, Ph.D., Principal Investigator — Laval University
Locations (1):
- Centre de recherche de l'Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Gilbert JA, Joanisse DR, Chaput JP, Miegueu P, Cianflone K, Almeras N, Tremblay A. Milk supplementation facilitates appetite control in obese women during weight loss: a randomised, single-blind, placebo-controlled trial. Br J Nutr. 2011 Jan;105(1):133-43. doi: 10.1017/S0007114510003119. PMID 21205360